CLINICAL TRIAL: NCT04356014
Title: Telangiectatic Palmoplantar Keratoderma in Systemic and Subacute Lupus Erythematosus : to a Form of Lichen Planus-like Lupus Erythematosus ?
Brief Title: Telangiectatic Palmoplantar Keratoderma in Systemic and Subacute Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0206
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-03

CONDITIONS: Systemic Lupus Erythematosus; Lichen Planus
Keywords: Palmoplantar keratoderma with livid telangiectatic erythema; Systemic lupus; Subacute lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lichen Planus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — paraffin-embedded and frozen cuteaneous biopsy specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Palmoplantar keratoderma (PPK) associated to livid telangiectatic erythema during systemic lupus erythematosus (SLE) and subacute cutaneous lupus erythematosus (SCLE) is a rare phenomenon seldom reported in literature. The investigators hypothesize that clinic-immunologic assessment and detailed investigation of cutaneous biopsy specimen of PPK and erythema of patients suffering from SLE and SCLE could lead to determine more precisely nosological settings of this injury. Report the different therapeutics with efficacy assessment could be helpful to highlight useful treatment for these patients.

DETAILED DESCRIPTION:
Context: Palmoplantar keratoderma (PPK) associated to livid telangiectatic erythema during systemic lupus erythematosus (SLE) is a rare phenomenon seldom reported in literature. To our knowledge no case has been described in subacute cutaneous lupus erythematosus (SCLE) so far. Pathogeny and etiologic origin are not clear: it could be no-specific cutaneous manifestation of SLE, verrucous chilblain lupus, lichen planus, discoid lupus erythematosus lesions, overlap syndrome or coexistence of both diseases.

Objective:

1. Determine clinical immunological and histopathological features of patients with PPK and livid telangiectatic erythema-associated suffering from SLE and SCLE
2. Describe the different therapeutics used and efficacy assessment Methods: Multicentric retrospective descriptive study reporting 14 patients with SLE or SCLE suffering from an acral livid erythematosus keratoderma, with clinical data regarding lupus erythematosus and acral keratoderma, immunological blood samples findings and histopathological results of keratoderma and livid erythema biopsies with direct immunofluorescence if performed. The treatments set down in order to heal are noted followed by efficacy assessment: total failure, partial remission, complete remission.

ELIGIBILITY:
Inclusion criteria:

* > 18 years old
* suffering from SLE or SCLE according to 2019 ACR/EULAR criteria
* With palmar and or plantar keratoderma with livid telangiectatic erythema

Exclusion criteria:

* < 18 years old
* suffering from lupus lesions without SLE or SCLE criteria
* without palmar and or plantar keratoderma with livid telangiectatic erythema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffering from SLE or SCLE with palmar and or plantar keratoderma with livid telangiectatic erythema
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Determine clinic immunologic features | 1 day
  Determine clinic immunologic features of patients with PPK and livid telangiectatic erythema-associated suffering from SLE and SCLE.
Determine clinic histopathologic features | 1 day
  Epidemiologic clinic immunologic histopathologic data

SECONDARY OUTCOMES:
Different therapeutics used | 1 day
  Describe the different therapeutics used. Report of the drug therapy used to heal acral keratoderma for each patient
Different therapeutics efficacy assessment | 1 day
  Efficacy assessment of the treatments: total failure, partial remission, complete remission

CONTACTS AND LOCATIONS:
Overall Officials: Didier BESSIS, PhD, Study Director — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC